CLINICAL TRIAL: NCT00657930
Title: Evaluation on Glycaemic Control and Weight Change of Once Daily Levemir® (Insulin Detemir) in Type 2 Diabetes Mellitus Treated by an Intensive Insulin Treatment (ICT)
Brief Title: Observational Study in Type 2 Diabetes Treated by an Intensive Insulin Treatment (ICT) Containing Once Daily Levemir® (Insulin Detemir)
Acronym: LEONCET2
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3526
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — observational study - dose and frequency to be prescribed by the physician as a result of standard clinical practice.
  Other Names: Levemir®

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to gain practical experience with once-daily Levemir administration in type 2 diabetes patients who were previously treated with Insulatard®, Humulin® N (NPH insulins) as basal insulin as part of their ICT under normal clinical practice conditions in Hungary.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic subjects on intensive insulin treatment (ICT)
* Eligibility for once daily insulin detemir administration
* Informed consent obtained before any observation-related activities

Exclusion Criteria:

* Known or suspected allergy to insulin detemir
* Subjects previously enrolled in the observation
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Type 2 Diabetes Mellitus patients on intensive insulin treatment
Sampling Method: Probability Sample
Enrollment: 2289 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficacy (HbA1c) | 24 weeks

SECONDARY OUTCOMES:
Body weight | 24 weeks
Hypoglycaemia frequency | 24 weeks
FBG variability | 24 weeks
Insulin dose change | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Budapest, Hungary

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com